CLINICAL TRIAL: NCT04565483
Title: Predictive Signature of Benralizumab Response
Acronym: BENRAPRED
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: AstraZeneca (Industry); Ministère de la Santé - France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC19_0292
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Asthma; Eosinophilic; Severe Asthma
Keywords: severe asthma; therapeutic monoclonal antibody; personalized medicine; transcriptomic; biomarkers
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BENRALIZUMAB (Experimental): Patients receive BENRALIZUMAB if they meet the criteria for inclusion and non-inclusion at the inclusion visit. Injections take place at the inclusion visit, at 1 month, 2 months, 4 months, 6 months, 8 months, 10 months and 12 months.
  Interventions: Drug: Benralizumab Prefilled Syringe

INTERVENTIONS:
Drug: Benralizumab Prefilled Syringe — Patients receive BENRALIZUMAB if they meet the criteria for inclusion and non-inclusion at the inclusion visit. Injections take place at the inclusion visit, at 1 month, 2 months, 4 months, 6 months, 8 months, 10 months and 12 months.
  Other Names: Transcriptomic

SUMMARY:
The objective of the study is to establish the predictive value of early blood gene expression signature of Benralizumab response associated with a significant reduction of the number of exacerbations in treated severe asthmatic patients.

This trial is a French, multicenter and no-randomized trial. Patients enrolled will be clinically followed for 16 months (the treatment period: 12 months and 1 month follow-up; 6 clinical visit on site and in phone call at 13 months)

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years old.
* Patients diagnosed with severe asthma (Chung and al, Eur Respir J 2014), i.e.:

  * asthma requiring high doses of ICS (>1000 microgram per day of Beclomethasone or equivalent) associated with LABA and/or systemic corticosteroids to be controlled over one year,
  * and/or uncontrolled asthma despite the later medications,
  * and/or a controlled asthma worsening after decreasing medications,
* Documented historical reversibility of FEV1 ≥12% and FEV1 gain ≥ 200 milliliter
* ACQ-7 score ≥ 1,5 at M0.
* ≥ 3 exacerbations in the 12 months prior to screening visit M-1.
* Eosinophil blood count ≥ 0,3 G/L at inclusion visit or in the 12 months prior to the inclusion visit. If eosinophil blood count is ≥ 0,15 G/L and < 0,3 G/L, an eosinophilic phenotype defined by at least 1 of the following criteria will be required:

  * Fractional Exhaled Nitric Oxide (FeNO) > 25 ppm at inclusion visit or in the 12 months prior to the inclusion visit.
  * Sputum eosinophils ≥ 3% at inclusion visit or in the 12 months prior to the inclusion visit.
* Patients who provide written informed consent prior to participation in the study

Exclusion Criteria:

* Patients diagnosed with difficult-to-treat asthma and/or with uncontrolled asthma differential diagnosis according to the judgment of the investigator (e.g., vocal cord dysfunction, gastroesophageal reflux disease, granulomatous eosinophilic vasculitis, obstructive sleep apnea syndrome, hyperventilation syndrome, allergic broncho-pulmonary aspergillosis, Carrington disease, DIPNECH, asthma/COPD overlap syndrome).
* Non-adherent patients to inhaled treatment (ICS + LABA).
* Active smokers or former smokers exceeding 20 packs year.
* Exacerbation at inclusion visit M0.
* Active malignancy or malignancy in remission over less than 5 years.
* Active parasitic infection or parasitic infection in the past 24 weeks.
* Hypersensitivity to Benralizumab or to any of the excipients of Fasenra® (histidine, histidine hydrochloride monohydrate, trehalose dihydrate, polysorbate 20)
* Patients requiring other immunosuppressive and immunomodulator drugs
* Patients requiring other biotherapy than Benralizumab, with or without French's marketing authorisation in severe asthma
* Patients requiring other biotherapy than Benralizumab that affects the immune system
* SARS-COV2 infection
* Pregnancy, lactation, or patients with childbearing potential refusing efficient contraceptive method.
* Patients under psychiatric condition altering their comprehension and their ability to give informed consent.
* Patients already enrolled in a clinical interventional research.
* Patients not affiliated to a health insurance plan
* Patients under guardianship, curators or safeguard of justice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Predictive value of early blood gene expression signature of Benralizumab | 12 months
  To establish the predictive value of early blood gene expression signature of Benralizumab response associated with a significant reduction of the number of exacerbations in treated severe asthmatic patients. We will evaluate an early blood gene expression signature of Benralizumab response through a clinically relevant reduction of the number of exacerbations at month 12 (M12).

SECONDARY OUTCOMES:
Molecular signature predictive of stabilization | 12 months
  To establish at M0 (baseline) a molecular signature predictive of stabilization in severe asthmatic patients treated by Benralizumab. At M0 a composite blood molecular signature predictive of reduction of the exacerbation rate at M12 in severe asthmatic patients treated by Benralizumab will be assessed. The definition of stable class of patients (low category) is used as a target for the prediction. The methods used for the primary objective are applied to secondary objective using similar input data on a different 3-class prediction target.
The stability of the signature over time | 0 month, 3 months, 6 months and 9 months
  To evaluate the stability of the signature over time (from early at M0, M3, to late prediction at M6 and M9) considering patient trajectories. The significance of center and the relevance of time dependent modelling will be evaluated using generalised mixed models on independently established molecular response signature. It is expected a robust and reproducible gene expression to assess the inter and intra-individual trajectories of the signature over time and across centers (from early at M0 and M3, to late prediction at M6 and M9).
The association of gene expression patterns | 12 months
  To evaluate the association of gene expression patterns with both objective and subjective improvement. Correlations network between blood gene expression of Benralizumab significant response will be assessed thanks to weighted gene correlation network analysis (gene co-expression network analysis (WGCNA)) with an expected increase in forced expiratory volume at one second (FEV1) + Asthma Quality of Life Questionnaire (AQLQ) + peak-flow values and expected decrease of Asthma Control Questionnaire-7 items (ACQ-7), -6 items (ACQ-6) scores.
Association of gene expression patterns and clinical characteristics | 0 months
  To evaluate association of gene expression patterns at M0 (baseline) and clinical characteristics of frequent exacerbations. Correlations network between blood gene expression at M0 and clinical characteristics of frequent exacerbations will be assessed thanks to WGCNA.
Stratification value of gene expression in severe asthma | 12 months
  To assess the stratification value of gene expression in severe asthma and its correlation with clinical subgroups and clinically meaningful variables such as number of exacerbations. Correlation network between stratification value of gene expressions in severe asthma and its correlation with clinical subgroups will be assessed thanks to WGCNA. This analysis is based on pairwise correlations between genetic variables and clinical variables underlying the amount of overall variance captured by high dimensional gene expression datasets.
Scenario-based cost-utility analysis | 12 months
  To conduct a scenario-based cost-utility analysis.Concerning cost-utility analysis, two strategies of treatment with Benralizumab will be compared: the first one will consider a strategy not using an early blood gene expression signature of Benralizumab response and the second will consider a simulated strategy using an early blood gene expression signature of Benralizumab response.

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Centre hospitalier Intercommunal Aix-en-Provence, Aix-en-Provence
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - Hôpital Bicêtre - AP-HP, Le Kremlin-Bicêtre
  - CH Mans, Le Mans
  - CHU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Assistance Publique des Hôpitaux de Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHR Orléans, Orléans
  - Hôpital Bichat - AP-HP, Paris
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - Hôpital FOCH, Suresnes
  - CHU Toulouse, Toulouse
  - Médipôle Hôpital Mutualiste de Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: Undecided